CLINICAL TRIAL: NCT05393128
Title: The Effect of Different Positions in Children After Cardiac Surgery On Vital Signs And Oxygen Saturation
Brief Title: The Effect of Different Positions in Children After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Principal Investigator Assist. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2021/21
Record Dates: First submitted 2022-03-02; First posted 2022-05-26 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Infant ALL
Keywords: pediatric heart surgery; position; infant
MeSH Terms: interventions — Control Groups; Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Supine position) (Other): The patient will remain in the supine position for 2 hours and will be followed up with the physician and nurse.
  After the patient is given one of the supine position, at any time during the 2-hour follow-up period, in case the patient's vital findings and SpO2 levels are beyond the normal findings, in case of a deterioration in the general condition related to the position or another reason, the position will be terminated with the physician's recommendation and the patient will be excluded from the sample. Or except these, in case the physician evaluates the patient and suggests that the position should be changed, the current position will be terminated, and the patient will be excluded from the sample by making a position change.
  Interventions: Procedure: Control group (Supine Position)
- Experimental Group (Right lateral position) (Experimental): The patient will remain in the right lateral position for 2 hours and will be followed up with the physician and nurse.
  After the patient is given one of the right lateral position, at any time during the 2-hour follow-up period, in case the patient's vital findings and SpO2 levels are beyond the normal findings, in case of a deterioration in the general condition related to the position or another reason, the position will be terminated with the physician's recommendation and the patient will be excluded from the sample. Or except these, in case the physician evaluates the patient and suggests that the position should be changed, the current position will be terminated, and the patient will be excluded from the sample by making a position change.
  Interventions: Procedure: Experimental Group (Right Lateral position)
- Experimental Group (Left lateral position) (Experimental): The patient will remain in the left lateral position for 2 hours and will be followed up with the physician and nurse.
  After the patient is given one of the left lateral position, at any time during the 2-hour follow-up period, in case the patient's vital findings and SpO2 levels are beyond the normal findings, in case of a deterioration in the general condition related to the position or another reason, the position will be terminated with the physician's recommendation and the patient will be excluded from the sample. Or except these, in case the physician evaluates the patient and suggests that the position should be changed, the current position will be terminated, and the patient will be excluded from the sample by making a position change.
  Interventions: Procedure: Experimental Group (Left Lateral position)

INTERVENTIONS:
Procedure: Control group (Supine Position) — In this group the patients will be given supine position.
  1. Body temperature, heart rate, respiration rate, blood pressure, oxygen saturation and CVP will be recorded before the process.
  2. The patient will be given supine position.
  3. The arms and the hands will be elevated and supported, the legs will be elevated and supported.
  4. The patient will be covered.
  5. The patient's vital signs, SpO2 levels will be registered right before giving position, on the 1st minute, on the 1st hour and on the 2nd hour from right after giving position.
  Arms: Control group (Supine position)
Procedure: Experimental Group (Right Lateral position) — In this group the patients will be given right lateral position.
  1. Body temperature, heart rate, respiration rate, blood pressure, oxygen saturation and CVP will be recorded before the process.
  2. The patient will be positioned supine and the bed will be straightened.
  3. Lines, probes will be taken to the right side of the patient and the patient will be turned with 60-90 degrees right lateral and the back will be supported with a pillow along the neck and sacrum.
  4. Between the legs will be supported with pillows.
  5. The patient's head will be elevated with 45-60 degrees.
  6. The patient will be covered :
  7. The patient's vital signs, SpO2 levels will be registered right before giving position, on the 1st minute, on the 1st hour and on the 2nd hour from right after giving position.
  Arms: Experimental Group (Right lateral position)
Procedure: Experimental Group (Left Lateral position) — In this group the patients will be given left lateral position.
  1. Body temperature, heart rate, respiration rate, blood pressure, oxygen saturation and CVP will be recorded before the process.
  2. The patient will be positioned supine and the bed will be straightened.
  3. Lines, probes will be taken to the left side of the patient and the patient will be turned with 60-90 degrees left lateral and the back will be supported with a pillow along the neck and sacrum.
  4. Between the legs will be supported with pillows.
  5. The patient's head will be elevated with 45-60 degrees.
  6. The patient will be covered :
  7. The patient's vital findings, SpO2 levels will be registered right before giving position, on the 1st minute, on the 1st hour and on the 2nd hour from right after giving position.
  Arms: Experimental Group (Left lateral position)

SUMMARY:
The objective of this study to determine the effects of giving right lateral, left lateral and supine positions on vital signs and oxygen saturation in children after cardiac surgery.

DETAILED DESCRIPTION:
Convenient ventilation management after pediatric cardiac surgery and the positioning of the patient helps to reduce the maximum intrathoracic pressure and venous stasis of the trunk and upper extremities that facilitates the drainage of the blood in the lungs. Due to the fact that the Pre-operative and post-operative management has tremendously changed for the last years, more detailed and up-to-date information is required related to the effect of the body position on the changes of the lung capacities and the pulmonary function. Based on this reason, this research was designed to determine the effect of three different positions as a randomized controlled prospective study.

In case the unit does not contain as routine any obstacle for position (unilateral oedema, ciculation disorder in the extremities, non-bilateral pulmonary atelectasis or dense infiltration, patients who cannot be administered dormicum or fentaver) right lateral, left lateral and supine positions are given. First positioning; also in routine, the standart position given to the first patients is supine position. The patient is first placed supine. Then his arms and legs are supported with support pillows. Transducer level and cuff pressure are controlled, SpO2 probe, ECG probes are controlled. If there's CVK connection, if there isn't any arterial connection, the cuff is controlled and in order to avoid heat loss the patient is covered after controling the body temperature and the position is completed.

In positioning, the 2nd method is right lateral positioning. In this positioning, the patient bed is straightened. Later on, the patient's SpO2 probe, ECG probes, CVK, arterial and cuff connections are once again moved to the right side of the patient and moved from below the patient's body without contact with the body in order to ensure the connections. Then, the patient is turned to right side with angle of 60 or 90 degrees and back is supported with a pillow from the neck to his sacrum, between the legs is also supported with a pillow. Afterwards, the patient's head is elevated with 45 to 60 degrees. Body temperature is controlled. The body is covered in order to avoid temperature loss and position is completed.

The third position that is used is left lateral position. In this positioning, the patient bed is straightened. Then, the patient's SpO2 probe, ECG probe, CVK, artery and cuff connections are transferred to the left side and the connections are made by passing the connections from below the pillow of the patient without touching the body. Later on, The patient is turned to left side with angle of 60 or 90 degrees to the left and the patient's back is supported with pillow from the neck until the sacrum, between the legs is again covered with a pillow. After that, the patient's head is elevated with 45-60 degrees. Body temperature is controlled, covered in order to avoid temperature loss and position is completed.

In this unit, after performing the applications related to the method used, the patient's vital signs and SpO2 are checked and recorded every half hour in the postoperative 24 hours, and hourly in the following processes.

In this study, implementation and data collection for each group will begin after the patient is admitted to the intensive care unit, after stabilization of the surgery (after the 12th hour). Until this time, the patient's follow-up is done in supine position. After stabilization, with the cooperation of the physician, it will continue to be supported by the right lateral and left lateral positions in addition to the supine position every 2 hours. Vital signs and SpO2 values of the patient will be recorded just before positioning, at the 1st minute, 1st hour and its 2nd hour after positioning.

ELIGIBILITY:
Inclusion Criteria:

* First time experiencing congenital cardiovascular surgery,
* Having Bilateral pulmonary atelectasis assessment,
* Not having any secondary congenital anomaly or chronic disease,
* Not having any neurologic symptoms,
* Being between 1 month - 1 year old
* Not having bilateral circulatory disorder and not having any obstacle to the position,
* Being Intubated
* Receiving 1 mg/kg dormicum, 0,1 mcg/kg fentaver infusion

Exclusion Criteria:

* Receiving Extra Corporal Membrane Exygenation support,
* Admitted to ICU with sternum exposed,
* Receiving Intraaortic balloon pump support,
* Being a Pre-op period patient,
* Having a non-bilateral circulatory disorder,
* Having unilateral thorax drain,
* Being extubated or being planned for extubation during the study period,
* Receiving Rocuranium,
* Not receiving Dormicum or fentaver

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Body Temperature | Data will be collected immediately before the position is given, at the 1st minute, at the 1st hour and at the 2nd hour after the position is given. The change in these time intervals will be assessed.
  This outcome will be considered as one of the vital signs. Body temperature measurement will be evaluated as axillary.
Change in Heart Rate | Data will be collected immediately before the position is given, at the 1st minute, at the 1st hour and at the 2nd hour after the position is given. The change in these time intervals will be assessed.
  Heart rate will be monitored.
Change in Blood Pressure | Data will be collected immediately before the position is given, at the 1st minute, at the 1st hour and at the 2nd hour after the position is given. The change in these time intervals will be assessed.
  Blood Pressure will be monitored.
Change in Respiratory Rate | Data will be collected immediately before the position is given, at the 1st minute, at the 1st hour and at the 2nd hour after the position is given. The change in these time intervals will be assessed.
  Respiratory rate will be monitored.
Change in Oxygen Saturation | Data will be collected immediately before the position is given, at the 1st minute, at the 1st hour and at the 2nd hour after the position is given. The change in these time intervals will be assessed.
  Oxygen Saturation will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Assist Prof, Principal Investigator — Acibadem University
Locations (1):
- Dr. Siyami Ersek Thoracic And Cardiovascular Surgery Education and Research Hospital, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silva ME, Feuser MR, Silva MP, Uhlig S, Parazzi PL, Rosa GJ, Schivinski CI. Pediatric cardiac surgery: what to expect from physiotherapeutic intervention? Rev Bras Cir Cardiovasc. 2011 Apr-Jun;26(2):264-72. doi: 10.1590/s0102-76382011000200018. English, Portuguese. PMID 21894418
- [Result] Thomas PJ, Paratz JD. Is there evidence to support the use of lateral positioning in intensive care? A systematic review. Anaesth Intensive Care. 2007 Apr;35(2):239-55. doi: 10.1177/0310057X0703500214. PMID 17444315
- [Result] de Laat E, Schoonhoven L, Grypdonck M, Verbeek A, de Graaf R, Pickkers P, van Achterberg T. Early postoperative 30 degrees lateral positioning after coronary artery surgery: influence on cardiac output. J Clin Nurs. 2007 Apr;16(4):654-61. doi: 10.1111/j.1365-2702.2006.01715.x. PMID 17402946
- [Result] Hickey PA, Pasquali SK, Gaynor JW, He X, Hill KD, Connor JA, Gauvreau K, Jacobs ML, Jacobs JP, Hirsch-Romano JC. Critical Care Nursing's Impact on Pediatric Patient Outcomes. Ann Thorac Surg. 2016 Oct;102(4):1375-80. doi: 10.1016/j.athoracsur.2016.03.019. Epub 2016 May 10. PMID 27173065